CLINICAL TRIAL: NCT04442620
Title: Prevention and Reversion of Non-Alcoholic Fatty Liver Disease in Obese Patients With Metabolic Syndrome by Mediterranean Diet and Physical Activity
Brief Title: Prevention and Reversion of NAFLD in Obese Patients With Metabolic Syndrome by Mediterranean Diet and Physical Activity
Acronym: FLIPAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Balearic Islands (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Josep1, Professor of Physiology, University of the Balearic Islands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201630.10
Record Dates: First submitted 2020-01-28; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Non Alcoholic Fatty Liver Disease; Metabolic syndrome; Mediterranean Diet; Physical activity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Motor Activity | interventions — Exercise; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1st group: Physical Activity and Mediterranean Diet (PA-MD) (Experimental): A first group of participants will be advised to reduce their caloric intake by 25-30% with a macronutrients distribution of 35-40% fat, 20% proteins, and 40-45% carbohydrates. Healthy fats (a maximum of 8-10% from saturated fats, >20% from monounsaturated fats, >10% from polyunsaturated fats and <300 mg/day of cholesterol) and low glycaemic index foods rich in fibre (not less than 30-35g /day) are strongly advised, together with foods rich in antioxidants, namely fruits and vegetables. Such diet reflects the traditional Mediterranean Diet described in the PREDIMED (Primary Prevention of Cardiovascular Disease with a Mediterranean Diet)-Plus study.
  As for physical activity, patients the participants will be recommended a 35 minutes interval training session three times a week. Physical activity sessions of 35 minutes will consist of 5 minutes warm-up, 20 minutes interval training, and 10 minutes breathing and stretching.
  Interventions: Other: Physical activity and Mediterranean Diet (PA-MD)
- 2nd group: High Meal Frequency of Mediterranean Diet (HMF-MD) (Experimental): A second group of participants will be advised to reduce their caloric intake by 25-30% with a macronutrients distribution of 30-35% fat, 25% proteins, and 40-45% carbohydrates. Healthy fats and low glycaemic index foods will be strongly advised, together with foods rich in antioxidants, namely fruits and vegetables. Participants will be advised to consume 7 meals a day, gradually reducing the caloric content at each main meal, and to walk 10.000 steps a day.
  Interventions: Other: High meal frequency of Mediterranean Diet (HMF-MD)
- 3rd group: Control diet (CD) (Active Comparator): A third group of participants will be advised to reduce their caloric intake by 25-30% with a macronutrients distribution of 30% fat, 15% proteins, and 55% carbohydrates, and maintain an adequate fibre (25g/day) and cholesterol (<250mg/day) intake. Meal frequency will be of 3-5 meals a day. Moreover, the participants will be advised to walk 10.000 steps a day.
  Interventions: Other: Control diet (CD)

INTERVENTIONS:
Other: Physical activity and Mediterranean Diet (PA-MD) — Physical Activity plus caloric restricted Mediterranean diet
  Arms: 1st group: Physical Activity and Mediterranean Diet (PA-MD)
Other: High meal frequency of Mediterranean Diet (HMF-MD) — High meal frequency of unaltered Mediterranean diet
  Arms: 2nd group: High Meal Frequency of Mediterranean Diet (HMF-MD)
Other: Control diet (CD) — Control Diet
  Arms: 3rd group: Control diet (CD)

SUMMARY:
This prospective randomized trial evaluates the role of customized dietary and physical activity intervention on the progression of Non-Alcoholic Fatty Liver Disease (NAFLD) in patients with obesity and presenting at least three of the main Metabolic Syndrome traits.

The project proposes a personalized nutritional intervention based on a Mediterranean customized diet which introduces plenty of antioxidant and anti-inflammatory bioactive components, coupled with physical activity promotion to prevent and reverse NAFLD among obese patients with metabolic syndrome. This will be compared with two more dietary strategies including a Mediterranean Diet intervention with seven meals a day and the conventional dietary approach proposed by the American Association for the Study of Liver Diseases (AASLD).

DETAILED DESCRIPTION:
There is currently no licensed pharmacological treatment for reversing Non-Alcoholic Fatty Liver Disease (NAFLD), this is why nutritional and lifestyle strategies are pivotal to ameliorate risk factors and prevent disease progression. Weight loss achieved by a weight loss diet and exercise is certainly the principal treatment for the amelioration of fatty liver, nevertheless quality of diet composition could also play a crucial role. Since oxidative stress and inflammation have been cited among the mechanisms involved in NAFLD, foods containing antioxidant and anti-inflammatory bioactive components should be considered when designing a nutritionally sound diet. The Mediterranean Diet, naturally rich in antioxidants and antinflammatory foods, together with personalised physical activity could have a variety of positive health effects, including the slowing down of degenerative diseases such as liver steatosis.

The present study aims to compare and evaluate the efficacy of three interventions on the pathophysiological mechanisms that may affect changes in liver fat deposits and progression of NAFLD in patients with obesity and presenting at least three of the main Metabolic Syndrome traits.

The first intervention group receives a caloric restricted Mediterranean Diet coupled with physical activity (delivered through guided gym classes); the second group receives a caloric restricted Mediterranean Diet distributed over 7 meals and advise to walk 10.000 steps a day; the third group receives the conventional diet proposed by the American Association for the Study of Liver Diseases (AASLD) and advise to walk 10.000 steps a day.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 60 years
* Diagnosis of NAFLD by ultrasound
* BMI ≥ 27 and < 40 kg/m2
* Meeting at least 3 of 5 criteria for the metabolic syndrome [as described in the International Diabetes Federation consensus]: (1) BMI >30kg/m² or increased waist circumference: ≥ 94 cm in males; ≥ 80 cm in females; (2) Triglycerides (TG) levels ≥ 150 mg/dL (1.7 mmol/L) or specific treatment; (3) Reduced HDL cholesterol: < 40 mg/dL (1.03 mmol/L) in males; < 50 mg/dL (1.29 mmol/L) in females or specific treatment; (4) Raised blood pressure: systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg or treatment of previously diagnosed hypertension; (5) Raised fasting plasma glucose (FPG) ≥ 100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes
* Written informed consent

Exclusion Criteria:

* Inability or unwillingness to give informed consent or communicate with staff study
* Documented history of prior cardiovascular disease [angina; myocardial infarction; coronary revascularization procedures; stroke (ischemic or hemorrhagic including transient ischemic attacks); symptomatic peripheral artery disease that required surgery or was diagnosed with vascular imaging techniques; ventricular arrhythmia; uncontrolled atrial fibrillation; congestive heart failure (New York Heart Association Class III or IV); hypertrophic myocardiopathy; and history of aortic aneurism >=5.5cm in diameter or aortic aneurism surgery]
* Documented history of prior liver diseases (other than NAFLD)
* Active cancer or a history of malignancy in the last 5 years
* Low predicted probability to change food habits according to the Stages of Change Model (Nigg, 1999)
* Unwillingness or inability to adhere to the dietary and physical activity intervention over the entire period of the study
* Failure to follow scheduled visits
* Weight loss (>5 kg) during 6 months prior to visit
* Previous surgical procedures for weight loss or scheduled bariatric surgery within the next 12 months
* Use of weight loss medications during 6 months prior to visit
* Previous history of bowel resection, inflammatory bowel disease
* Obesity associated with endocrine disease (except treated hypothyroidism)
* Allergy to Mediterranean diet foods or components
* Severe psychiatric disorders (schizophrenia, bipolar disorder, eating disorders, or depression with hospitalization within the last 6 months) or Beck Depression Inventory score > 30
* Severe condition with less than 24 months life expectancy
* Chronic abuse of drugs or alcohol (>21 and >14 units of alcohol a week for men and women, respectively; 1 unit = 125 mL of wine)
* Treatment with steroids
* Pregnancy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in liver steatosis | At baseline, 6, 12 and 24 months
  The primary outcome is to measure the change of liver steatosis (expressed as percentage of liver steatosis) after applying a different intervention to each group (PA-MD; HMF-MD; or CD) of participants with metabolic syndrome.
  It will be measured (at baseline, and after 6, 12 and 24 months of intervention) by means of a 1.5-T Magnetic Resonance Imaging (MRI) (Signa Explorer 1.5T, General Electric Healthcare, Chicago, Illinois., U.S.A) by using a 12-channel phased-array coil.

SECONDARY OUTCOMES:
Changes in liver fibrosis | At baseline, 6, 12 and 24 months
  The secondary otucome is to measure the changes of liver fibrosis (expressed as percentage of liver fibrosis) after applying a different intervention to each group (PA-MD; HMF-MD; or CD) of participants with metabolic syndrome.
  It will be measured (at baseline, and after 6, 12 and 24 months of intervention) by using Shear Wave Measurement (SWM) (Hitachi Ltd, Japan) and the echograph Arietta V70 (Hitachi Medical System Europe Holding AG, Steinhausen, Switzerland).

CONTACTS AND LOCATIONS:
Overall Officials: Josep A Tur, PhD, Principal Investigator — University of the Balearic Islands
Locations (1):
- University of the Balearic Islands, Palma, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No
There are restrictions on the availability of data for the FLIPAN trial, due to the signed consent agreements around data sharing, which only allow access to external researchers for studies following the project purposes. Requestors wishing to access the FLIPAN trial data used in this study can make a request to the FLIPAN trial. Steering Committee chair: pep.tur@uib.es. The request will then be passed to members of the FLIPAN Steering Committee for deliberation.

REFERENCES:
- [Derived] Quetglas-Llabres MM, Monserrat-Mesquida M, Bouzas C, Llompart I, Mateos D, Casares M, Ugarriza L, Martinez JA, Tur JA, Sureda A. Mediterranean Diet Improves Plasma Biomarkers Related to Oxidative Stress and Inflammatory Process in Patients with Non-Alcoholic Fatty Liver Disease. Antioxidants (Basel). 2023 Mar 29;12(4):833. doi: 10.3390/antiox12040833. PMID 37107208